CLINICAL TRIAL: NCT00199056
Title: Multicenter Trial for Treatment of Acute Lymphocytic Leukemia in Adults (Pilot Study 06/99)
Brief Title: German Multicenter Trial for Treatment of Newly Diagnosed Acute Lymphoblastic Leukemia in Adults (06/99)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Head of GMALL, Goethe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMALL10
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Adult Acute Lymphocytic Leukemia
Keywords: ALL; Treatment; De Novo; Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dexamethasone; Prednisolone; Cyclophosphamide; Methotrexate; Vincristine; Vindesine; Daunorubicin; Asparaginase; Granulocyte Colony-Stimulating Factor; Cytarabine; Mercaptopurine; Etoposide; Doxorubicin; Thioguanine; Teniposide; Idarubicin; fludarabine; Ifosfamide; Stem Cell Transplantation

INTERVENTIONS:
Drug: Dexamethasone / Prednisolone
Drug: Cyclophosphamide
Drug: Methotrexate
Drug: Vincristine / Vindesine
Drug: Daunorubicin
Drug: Asparaginase
Drug: G-CSF
Drug: Cytarabine
Drug: 6-Mercaptopurine
Drug: VP16
Drug: Adriamycin
Drug: Thioguanine
Drug: VM26
Drug: Idarubicin
Drug: Fludarabine
Drug: Ifosfamide
Procedure: CNS irradiation
Procedure: Mediastinal irradiation (if residual tumor)
Procedure: stem cell transplantation

SUMMARY:
The study evaluates the efficacy and tolerability of an intensified induction and consolidation therapy. Thereafter patients receive individualised treatment stratified according to relapse risk with stem cell transplantation for patients with high and very high risk of relapse. Patients with standard risk receive further consolidation and reinduction chemotherapy. In parallel minimal residual disease (MRD) is evaluated. A MRD based risk stratification and treatment decision is developed.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia (pro-B, common, pre-B, early T, T)
* Age 15-65 yrs (*55-65 years if biologically younger according to general condition)

Exclusion Criteria:

* Severe comorbidity
* Cytostatic pre-treatment
* Pregnancy
* Missing written informed consent

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225
Dates: Start 1999-10 (Actual); Primary Completion 2003-11 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Remission rate,Remission duration,Disease free survival,Overall survival

SECONDARY OUTCOMES:
Time and dose compliance,Realisation of SCT,Toxicity according to WHO,Course of MRD

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD,PhD, Study Chair — University Hospital Frankfurt, Medical Dept. II
Locations (1):
- University Hospital, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- [Derived] Kobitzsch B, Gokbuget N, Schwartz S, Reinhardt R, Bruggemann M, Viardot A, Wasch R, Starck M, Thiel E, Hoelzer D, Burmeister T. Loss-of-function but not dominant-negative intragenic IKZF1 deletions are associated with an adverse prognosis in adult BCR-ABL-negative acute lymphoblastic leukemia. Haematologica. 2017 Oct;102(10):1739-1747. doi: 10.3324/haematol.2016.161273. Epub 2017 Jul 27. PMID 28751559
- [Derived] Herold T, Schneider S, Metzeler KH, Neumann M, Hartmann L, Roberts KG, Konstandin NP, Greif PA, Braundl K, Ksienzyk B, Huk N, Schneider I, Zellmeier E, Jurinovic V, Mansmann U, Hiddemann W, Mullighan CG, Bohlander SK, Spiekermann K, Hoelzer D, Bruggemann M, Baldus CD, Dreyling M, Gokbuget N. Adults with Philadelphia chromosome-like acute lymphoblastic leukemia frequently have IGH-CRLF2 and JAK2 mutations, persistence of minimal residual disease and poor prognosis. Haematologica. 2017 Jan;102(1):130-138. doi: 10.3324/haematol.2015.136366. Epub 2016 Aug 25. PMID 27561722
- [Derived] Gokbuget N, Stanze D, Beck J, Diedrich H, Horst HA, Huttmann A, Kobbe G, Kreuzer KA, Leimer L, Reichle A, Schaich M, Schwartz S, Serve H, Starck M, Stelljes M, Stuhlmann R, Viardot A, Wendelin K, Freund M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Outcome of relapsed adult lymphoblastic leukemia depends on response to salvage chemotherapy, prognostic factors, and performance of stem cell transplantation. Blood. 2012 Sep 6;120(10):2032-41. doi: 10.1182/blood-2011-12-399287. Epub 2012 Apr 4. PMID 22493293
- [Derived] Gokbuget N, Kneba M, Raff T, Trautmann H, Bartram CR, Arnold R, Fietkau R, Freund M, Ganser A, Ludwig WD, Maschmeyer G, Rieder H, Schwartz S, Serve H, Thiel E, Bruggemann M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Adult patients with acute lymphoblastic leukemia and molecular failure display a poor prognosis and are candidates for stem cell transplantation and targeted therapies. Blood. 2012 Aug 30;120(9):1868-76. doi: 10.1182/blood-2011-09-377713. Epub 2012 Mar 22. PMID 22442346
- [Derived] Burmeister T, Meyer C, Schwartz S, Hofmann J, Molkentin M, Kowarz E, Schneider B, Raff T, Reinhardt R, Gokbuget N, Hoelzer D, Thiel E, Marschalek R. The MLL recombinome of adult CD10-negative B-cell precursor acute lymphoblastic leukemia: results from the GMALL study group. Blood. 2009 Apr 23;113(17):4011-5. doi: 10.1182/blood-2008-10-183483. Epub 2009 Jan 14. PMID 19144982
- See also: German Leukemia Trial Registry — http://www.studienregister-online.de